CLINICAL TRIAL: NCT06605417
Title: Understanding the Transition from Normal Melanocytes to Nevus to Melanoma (NevustoMel)
Brief Title: Understanding the Transition from Normal Melanocytes to Nevus to Melanoma
Acronym: NevustoMel
Status: Recruiting | Type: Observational
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Institut National de la SantÃ© Et de la Recherche MÃ©dicale, France (Unknown); University Hospital Tuebingen (Other); University of Florence (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); University Of Perugia (Other); German Cancer Research Center (Other); Karolinska Institutet (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Institut Curie (Other); Medical University of Gdansk (Other); Princess Maxima Center for Pediatric Oncology (Other); Institut Català d'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2023/0843; HORIZON-MISS-2021-CANCER-02-03 (Other Grant/Funding Number: European Comission)
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-09

CONDITIONS: Congenital Melanocytic Nevi; Melanoma, Skin; Nevi and Melanomas
Keywords: Congenital melanocytic nevi; Melanoma; Liquid biopsy; cfDNA; Methylomics; L/GCMN; RNAseq; Molecular profiles
MeSH Terms: conditions — Melanoma; Nevi and Melanomas | interventions — Sequence Analysis, RNA; Liquid Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — * Cell-free DNA will be extracted from patient's blood and saliva.
  * DNA and RNA extracted from Formalin-Fixed Paraffin-Embedded (FFPE) patient tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- L/GCMN: Patients with congenital nevus with estimated size of 20 cm or more in adulthood (> 18 years old)
  Interventions: Genetic: Methylomics; Genetic: RNA sequencing; Genetic: Spatial transcriptomics; Genetic: Liquid biopsy
- Melanoma: Patients affected with Spitz-type or conventional melanomas in patients under 30 years of age
  Interventions: Genetic: Methylomics; Genetic: RNA sequencing; Genetic: Spatial transcriptomics; Genetic: Liquid biopsy

INTERVENTIONS:
Genetic: Methylomics — Methylomics analysis of FFPE blocks and frozen tissues
Genetic: RNA sequencing — RNA sequencing of FFPE blocks and frozen tissues
Genetic: Spatial transcriptomics — Spatial transcriptomics of FFPE blocks and frozen tissues
Genetic: Liquid biopsy — cfDNA characterization extracted from blood/saliva

SUMMARY:
The primary objective of this study is to identify the molecular identity profiles of all cellular states that characterize the progression from benign nevi to malignant melanoma in CAYA patients with L/GCMN. The secondary objectives are:

* To longitudinally characterize the cell-free DNA (cfDNA) from CAYA patients.
* To improve the early diagnosis and treatments for intermediate conditions such as L/GCMN through evidence-based interpretation of personal risk from endogenous or exogenous sources.
* To test pre-clinical strategies to best model and improve patient response.

DETAILED DESCRIPTION:
NevustoMel is an international multicentric retrospective cohort study with molecular and experimental design. It will involve the genomic characterization of cell-free DNA and affected tissues from patients. Methylomics and single-cell multi-omics will be used to identify co-existing molecular (transcriptional and epigenomic) states at single-cell level and will be generated from affected tissues. These results will be exploited using machine learning-assisted integration of multi-modal transcriptomics, epigenomics and spatial information. Integrated analyses of single-nucleus RNA sequencing from a selection of frozen tissues and spatial transcriptomics on formalin-fixed paraffin-embedded samples will allow the comparison of the findings to ground-state Human Developmental Cell Atlas data. Distinctions will be validated either with in situ hybridization (such as RNA sequencing) or immunostaining on test cohort tissues. These results will be complemented with in vitro functional analyses, high throughput sequencing and bioinformatic analyses.

ELIGIBILITY:
Inclusion criteria:

* Congenital nevus with estimated size of 20 cm
* Be over 18 years of age

Exclusion criteria:

* No available biological material
* Not having signed the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Review and/or analysis of pre-existing medical records, biological samples and data collected from patients that have been visited at the different participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Molecular identity profiles | 26 months
  Molecular identity profiles of all cellular states that characterize the progression from benign nevi to malignant melanoma in children, adolescents and young adults (CAYA) patients with large/giant congenital melanocytic nevi (L/GCMN)

SECONDARY OUTCOMES:
cfDNA profiles | 26 months
  Longitudinal characterization of the cell-free DNA (cfDNA) of CAYA patients
Improve the early diagnosis and treatment of L/GCMN | 26 months
  Improve the early diagnosis and treatments for intermediate conditions such as L/GCMN through evidence-based interpretation of personal risk from endogenous or exogenous sources.
Test pre-clinical strategies for L/GCMN | 26 months
  Test pre-clinical strategies to best model and improve patient response with intermediate lesions such as L/GCMN

CONTACTS AND LOCATIONS:
Locations (2):
- French National Institute of Health and Medical Research, Marseille, France
- Hospital Clínic de Barcelona (Dermatology service), Barcelona, Spain